CLINICAL TRIAL: NCT02205996
Title: The Effects of Hypoglycaemia on Platelets Function and Inflammatory Markers in People With Type 2 Diabetes and Normal Controls.
Brief Title: The Effects of Hypoglycaemia in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Thozhukat Sathyapalan, Dr, University of Hull
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11/YH/0161
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Hypoglycaemia; Platelets; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Inflammation | interventions — Insulin; Insulin, Regular, Human; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controls (Active Comparator): Weight-matched healthy controls. Euglycaemic Hypoglycaemic insulin clamp. Using hyperinsulinaemic clamps, blood glucose levels were stabilised over 1 hour to reach 5 mmol/L and maintained at that level for 1 hour, then gradually reduced over 1 hour to 2.8 mmol/L and maintained at that level for 1 hour. Blood samples were collected at times 0 (baseline), 2 hours (euglycaemia), 4 hours (hypoglycaemia) and at 24 hours after the clamp studies.
  Interventions: Drug: Insulin (Humulin S); Device: Euglycaemic Hypoglycaemic Insulin clamp
- Type 2 diabetes (Active Comparator): People with a known diagnosis of type 2 diabetes. Euglycaemic Hypoglycaemic Insulin clamp. Using hyperinsulinaemic clamps, blood glucose levels were stabilised over 1 hour to reach 5 mmol/L and maintained at that level for 1 hour, then gradually reduced over 1 hour to 2.8 mmol/L and maintained at that level for 1 hour. Blood samples were collected at times 0 (baseline), 2 hours (euglycaemia), 4 hours (hypoglycaemia) and at 24 hours after the clamp studies.
  Interventions: Drug: Insulin (Humulin S); Device: Euglycaemic Hypoglycaemic Insulin clamp

INTERVENTIONS:
Drug: Insulin (Humulin S) — Using insulin and glucose infusions (hyperinsulinaemic clamps), blood glucose levels were stabilised over 1 hour to reach 5 mmol/L and maintained at that level for 1 hour, then gradually reduced over 1 hour to 2.8 mmol/L and maintained at that level for 1 hour. Blood samples were collected at times 0 (baseline), 2 hours (euglycaemia), 4 hours (hypoglycaemia) and at 24 hours after the clamp studies.
  Other Names: Glucose (20% Dextrose).
Device: Euglycaemic Hypoglycaemic Insulin clamp

SUMMARY:
Strict glycaemic control has been associated with increased hypoglycaemia and mortality rate, the cause of which was unclear, in subjects with type 2 diabetes. In this study, we hypothesised that acute hypoglycaemia will result in platelet activation in people with type 2 diabetes to a higher degree than controls.

DETAILED DESCRIPTION:
Type 2 diabetes is associated with increased risk of cardiovascular disease. Although the United Kingdom Prospective Diabetes Study (UKPDS) follow-up data suggested reduced macrovascular complications with tight glycaemic control, recent studies in people with type 2 diabetes failed to replicate these findings. Furthermore, all-cause mortality was found to be increased with strict glycaemic control in the Action to Control Cardiovascular Risk in Diabetes (ACCORD) study. The cause of the increased deaths remains unclear.

Strict glycaemic control is associated with increased risk of hypoglycaemia. Although, hypoglycaemia has traditionally been considered a complication of the treatment for type 1 diabetes, it has recently been recognised as a problem in people with type 2 diabetes particularly those on insulin therapy. In the ACCORD study, the risk of death was significantly increased in those with one or more episode of severe hypoglycaemia in both the strict and standard study treatment arms. As plasma glucose falls to below 4.0 mmol/L, a series of defence mechanisms occur, at an individualised glycaemic thresholds, to reverse hypoglycaemia including a rise in catecholamine levels. This may lead to hypokalaemia, prolonged QT interval, and cardiac arrhythmias. It may also lead to impaired cardiovascular autonomic function for up to 16 hours afterwards; increased inflammatory markers; platelet activation and promote vascular damage. As the majority of studies assessing the effects of hypoglycaemia on cardiovascular risk markers are conducted in people with type 1 diabetes and healthy controls, their findings may not necessarily be applicable to people with type 2 diabetes. In particular, the effects of hypoglycaemia on platelet function and thrombotic risk in people with type 2 diabetes require further clarification. In this study, we hypothesised that acute hypoglycaemia will result in platelet activation in people with type 2 diabetes to a higher degree than controls.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers:

   * Males or females
   * On no medications except for the contraceptive pill and without medical illnesses in the last three months.
   * Non-smokers
   * 40 - 60 years of age.
2. T2DM subjects:

   * Males or females
   * Diagnosis of T2DM
   * 40 - 60 years of age
   * HbA1C: 6.5 - 9.5%
   * Duration of diabetes 1 - 10 years
   * Diabetes treated with diet, or tablets only.

Exclusion Criteria:

1. Healthy volunteers:

   * Pregnancy
   * Lack of contraception in women of child bearing age
   * Chronic medical conditions
   * Current smokers
   * Evidence of ischaemia on ECG
   * Drop attacks
   * Alcohol or drug abuse
   * Psychiatric illness
   * Previous history of seizure
   * Alcohol or drug abuse
2. Type 2 diabetes subjects:

   * Pregnancy
   * Current smokers
   * Recurrent episodes of hypoglycaemia
   * Treatment with anti-platelet or anti-coagulation therapy
   * History of ischaemic heart disease, stroke or peripheral vascular disease
   * Epilepsy
   * Drop attacks
   * Evidence of ischaemia on ECG
   * Insulin treated T2DM
   * History of microvascular disease (retinopathy, nephropathy or neuropathy).
   * Alcohol or drug abuse
   * Psychiatric illness

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To examine the effect of hypoglycaemia on platelet surface expression of platelet activation markers P-selectin and fibrinogen binding. | Up to 24 hours after euglycaemic hypoglycaemic clamp
  Platelet surface expression of activation markers, P-selectin and fibrinogen binding, were measured in the resting state (unstimulated samples) and in response to stimulation with platelet agonist adenosine diphosphate, and platelet inhibitor prostacyclin.
  A change in platelet function from times 0 (baseline), to 2 hours (euglycaemia), 4 hours (hypoglycaemia) and 24 hours after the clamp studies was measured and compared between the two groups.

SECONDARY OUTCOMES:
To measure changes in markers of inflammation (high sensitivity C-reactive protein) and endothelial function using EndoPat 2000 | Up to 24h after euglycaemic hypoglycaemic clamp
  High sensitivity C-reactive protein was measured at baseline (time 0), 2 hours (euglycaemia), 4 hours (hypoglycaemia) and 24 hours after clamp studies. Changes from baseline were compared between the groups.
  EndoPat was measured before the insulin clamp and 24 hours afterwards and changes were compared between the two groups.

OTHER OUTCOMES:
To assess the effects of hypoglycaemia on participants scores on cognitive function tests | Up to 24h after euglycaemic hypoglycaemic clamp
  Three cognitive function tests (Tower of Hanoi; Dual Task test and The Digit symbol-coding) were measured at baseline (time 0), 2 hours (euglycaemia), 4 hours (hypoglycaemia) and 24 hours after insulin clamp studies. Changes from baseline in each of these tests in response to the insulin clamp were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Atkin, PhD, Principal Investigator — Hull York Medical School
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom

REFERENCES:
- [Derived] Moin ASM, Sathyapalan T, Atkin SL, Butler AE. The severity and duration of Hypoglycemia affect platelet-derived protein responses in Caucasians. Cardiovasc Diabetol. 2022 Oct 6;21(1):202. doi: 10.1186/s12933-022-01639-w. PMID 36203210
- [Derived] Moin ASM, Nandakumar M, Kahal H, Sathyapalan T, Atkin SL, Butler AE. Heat Shock-Related Protein Responses and Inflammatory Protein Changes Are Associated with Mild Prolonged Hypoglycemia. Cells. 2021 Nov 10;10(11):3109. doi: 10.3390/cells10113109. PMID 34831332
- [Derived] Moin ASM, Kahal H, Al-Qaissi A, Kumar N, Sathyapalan T, Atkin SL, Butler AE. Amyloid-related protein changes associated with dementia differ according to severity of hypoglycemia. BMJ Open Diabetes Res Care. 2021 Apr;9(1):e002211. doi: 10.1136/bmjdrc-2021-002211. PMID 33931404